CLINICAL TRIAL: NCT02604563
Title: Aging, Geriatric Syndromes and Clonal Hematopoiesis
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Edward P. Evans Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 201511019
Record Dates: First submitted 2015-11-09; First posted 2015-11-13 (Estimated); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Geriatrics; Aged; Geriatric Syndromes; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Mental Status and Dementia Tests; Walking Speed; Hand Strength; Body Height; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Peripheral blood
  * Buccal swab or tongue brushing
  * Optional bone marrow biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Arm A: Clonal hematopoiesis: * Complete several self-administered health assessments at baseline and every 6 months until death.
  * Cognitive assessment, Gait Speed, grip strength, blood pressure, height, and weight will be performed by a member of the research team at baseline and every 6 months until death.
  * Peripheral blood draw will occur at baseline and no more than every 6 months until death.
  * Buccal swabs will occur at baseline and repeated as necessary, but not more than every 6 months until death
  * May be approached about optional bone marrow biopsy
  Interventions: Other: Cognitive Assessment; Other: Activities of Daily Living Questionnaire; Other: Instrumental Activities of Daily Living, subscale of the OARS; Other: Karnofsky Self-reported Performance Rating Scale; Other: Number of Falls; Other: Physical Health Section, subscale of the OARS; Other: MOS Social Activity Survey; Other: Unintentional Weight Loss; Genetic: Peripheral Blood Draw; Genetic: Buccal Swab; Other: Heart Health and Smoking History from BRFSS questionnaire; Other: Gait Speed; Other: Grip Strength; Other: Height and Weight measurements; Other: Blood pressure measurement; Procedure: Optional bone marrow biopsy
- Arm B: No clonal hematopoiesis: * Complete several self-administered health assessments at baseline and every 6 months until death.
  * Cognitive assessment, Gait Speed, grip strength, blood pressure, height, and weight will be performed by a member of the research team at baseline and every 6 months until death.
  * Peripheral blood draw will occur at baseline and no more than every 6 months until death.
  * Buccal swabs will occur at baseline and repeated as necessary, but not more than every 6 months until death
  * May be approached about optional bone marrow biopsy
  Interventions: Other: Cognitive Assessment; Other: Activities of Daily Living Questionnaire; Other: Instrumental Activities of Daily Living, subscale of the OARS; Other: Karnofsky Self-reported Performance Rating Scale; Other: Number of Falls; Other: Physical Health Section, subscale of the OARS; Other: MOS Social Activity Survey; Other: Unintentional Weight Loss; Genetic: Peripheral Blood Draw; Genetic: Buccal Swab; Other: Heart Health and Smoking History from BRFSS questionnaire; Other: Gait Speed; Other: Grip Strength; Other: Height and Weight measurements; Other: Blood pressure measurement; Procedure: Optional bone marrow biopsy
- Arm C: No clonal hematopoiesis & no follow-up: * Complete several self-administered health assessments at baseline with no further follow-up
  * Cognitive assessment, Gait Speed, grip strength, blood pressure, height, and weight will be performed by a member of the research team at baseline with no further follow-up
  * Peripheral blood draw will occur at baseline with no further follow-up
  * Buccal swabs will occur at baseline with no further follow-up
  Interventions: Other: Cognitive Assessment; Other: Activities of Daily Living Questionnaire; Other: Instrumental Activities of Daily Living, subscale of the OARS; Other: Karnofsky Self-reported Performance Rating Scale; Other: Number of Falls; Other: Physical Health Section, subscale of the OARS; Other: MOS Social Activity Survey; Other: Unintentional Weight Loss; Genetic: Peripheral Blood Draw; Genetic: Buccal Swab; Other: Heart Health and Smoking History from BRFSS questionnaire; Other: Gait Speed; Other: Grip Strength; Other: Height and Weight measurements; Other: Blood pressure measurement
- Arm D: Hip replacement: * Complete several self-administered health assessments at baseline and every 6 months until death.
  * Cognitive assessment, Gait Speed, grip strength, blood pressure, height, and weight will be performed by a member of the research team at baseline and every 6 months until death.
  * Participants with or without clonal hematopoiesis who are undergoing hip replacement
  * Peripheral blood draw will occur at baseline and no more than every 6 months until death.
  * Buccal swabs will occur at baseline and repeated as necessary, but not more than every 6 months until death
  * May be approached about optional bone marrow biopsy
- Arm E: Trauma: -Blood sample at the time of admission with initial bloodwork. For inpatient participants, weekly follow-up samples will be drawn with morning phlebotomy. A follow-up sample collection will occur 4-7 weeks after discharge.
  Interventions: Procedure: Blood draw for trauma measurements

INTERVENTIONS:
Other: Cognitive Assessment — -Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Activities of Daily Living Questionnaire — * 10 items about daily functional status
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Instrumental Activities of Daily Living, subscale of the OARS — * 7 items about daily functional status
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Karnofsky Self-reported Performance Rating Scale — * 1 item about daily functional status
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Number of Falls — * 1 item about daily functional status
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Physical Health Section, subscale of the OARS — * 13 items about comorbidity
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: MOS Social Activity Survey — * 4 items about social activity
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Unintentional Weight Loss — * 2 items about nutrition
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Genetic: Peripheral Blood Draw — -Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Genetic: Buccal Swab — * Participants will rinse their mouths 2 times with water for 20-30 seconds and discard the expectorated sample. One side of the inner cheek (buccal mucosa) will then be scraped with a cotton swab 20 times (alternatively, the tongue will be brushed 20 times with a toothbrush)
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Heart Health and Smoking History from BRFSS questionnaire — * 7 items about heart health and smoking history
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Gait Speed — * Research coordinator will test gait speed
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Grip Strength — * Research coordinator will test grip strength
  * Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Height and Weight measurements — -Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Other: Blood pressure measurement — -Baseline and no more frequently than every 6 months until death
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis; Arm C: No clonal hematopoiesis & no follow-up
Procedure: Optional bone marrow biopsy — -1 optional bone marrow biopsy
  Groups: Arm A: Clonal hematopoiesis; Arm B: No clonal hematopoiesis
Procedure: Blood draw for trauma measurements — -For Arm E only
  Groups: Arm E: Trauma

SUMMARY:
In this study the investigators will incorporate a wide range of clinical variables associated with aging and cardiovascular disease to determine whether they are associated with mutation status independent of chronologic age. Clinically, aging can be operationalized using geriatric assessment, which entails a comprehensive multi-dimensional assessment of the health of an older adult, including measures of comorbidity, polypharmacy, functional status, cognition, depression, falls, social activities and social support. Given that aging is heterogeneous, geriatric assessment allows greater specificity for aging than chronological age alone.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years of age.
* Able to understand written and spoken English.
* Able to understand and willing to sign an IRB-approved written informed consent document (or that of a legally authorized representative, if applicable for the trauma cohort)

Exclusion Criteria:

* Inability or unwillingness to complete health questionnaire.
* History of a recent (<30 days) acute viral illness.
* Current cancer diagnosis and currently receiving chemotherapy or undergoing radiation therapy. A prior history of cancer is allowed if the participant completed therapy > 1 year prior to enrollment; participants with a prior diagnosis of cancer will be asked to sign a release of information for the research team to obtain records regarding their prior cancer treatment.
* Current use of drugs that cause DNA damage (e.g. Cytoxan, azathioprine, etc.) for the treatment of a non-malignant disease.
* Vulnerable populations (e.g. prisoners).
* Known infection with Hepatitis B or C, HTLV, or HIV.
* Additional exclusion for optional bone marrow aspirate/biopsy substudy:

  * Use of medications for anticoagulation or "blood thinning" including warfarin, low molecular weight heparins (enoxaparin, daltaparin) or direct-acting oral anticoagulants (dabigatran, rivaroxaban, apixaban, edoxaban or betrixaban)
  * allergy to lidocaine or other local anesthetics.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants seen in Washington University School of Medicine clinics.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-03-10 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Background mutation rate in hematopoietic stem cells from older adults regardless of a prior cancer diagnosis as measured by the number and frequency of hematopoietic-specific mutations | Estimated to be 10 years
  -The investigators will sequence the coding region of some or all of the genes in an individual's blood cells and compare results to their matched mouth cells to define hematopoietic-specific mutations. The number of hematopoietic-specific mutations per individual and the frequency of individuals with mutations will be measured.
Presence or absence of geriatric syndromes as measured by hematopoietic stem cell mutations | Estimated to be 10 years
  -The presence or absence of geriatric syndromes will be correlated with the mutation status of individuals.
Determine the natural history of mutations in older adults with clonal hematopoiesis as measured by risk to develop blood cancer/geriatric syndrome/illness/cardiovascular disease | Estimated to be 10 years
  -Individuals with mutations will be followed longitudinally to monitor the fraction of hematopoietic cells with mutations, the functional consequences of mutations in their blood cells, and the risk of developing a blood cancer, geriatric syndrome, cardiovascular disease, or other illness.
Presence or absence of cardiovascular disease as measured by hematopoietic stem call mutations | Estimated to be 10 years
Determine whether expansion of clonal hematopoiesis (CH) occurs following acute trauma | Estimated to be 10 years
  -Measures change in variant allele fraction

CONTACTS AND LOCATIONS:
Overall Officials: Meagan Jacoby, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu